CLINICAL TRIAL: NCT03940612
Title: Use of Probiotic for the Prevention of Re-occurrence Vaginal Candidiasis in Pregnant Women
Brief Title: Probiotic for Vaginal Candidiasis in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: SYNBIO TECH INC. Kaohsiung Taiwan (Unknown)
Responsible Party: Principal Investigator, Min-Tze LIONG, Prof. Dr., Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: USM/JEPeM/18090421
Record Dates: First submitted 2019-04-17; First posted 2019-05-07 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Vaginal Diseases
Keywords: candidiasis; probiotic; STP4; pregnant
MeSH Terms: conditions — Vaginal Diseases; Candidiasis | interventions — Pharmaceutical Preparations; Probiotics

STUDY DESIGN:
Intervention Model Description: Placebo and STP4 will be administered via a parallel design
Who Masked: Participant, Care Provider, Investigator
Masking Description: Masking will be subjected to Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STP4 (product with probiotics) (Experimental): Dietary Supplement: STP4
  Interventions: Dietary Supplement: STP4 (product with probiotics)
- Placebo (product without probiotics) (Experimental): Dietary Supplement: Placebo
  Interventions: Dietary Supplement: Placebo (product without probiotics)

INTERVENTIONS:
Dietary Supplement: STP4 (product with probiotics) — STP4 contains Lactobacillus plantarum LP115, Lactobacillus helveticus LA25, Lactobacillus rhamnosus LRH10, Lactobacillus paracasei LPC12, Lactobacillus fermentum LF26, Lactobacillus delbrueckii subsp. lactis, LDL114. Administration at 10 log CFU/day for 8-weeks.
  Arms: STP4 (product with probiotics)
Dietary Supplement: Placebo (product without probiotics) — Capsules are similar to STP4 except the presence of probiotics. Administration daily for 8-weeks.
  Arms: Placebo (product without probiotics)

SUMMARY:
This project aims to study the benefits of a probiotic product, STP4 for vaginal health properties, primarily prevention of vaginal candidiasis, among pregnant women in second and third trimester pregnancy.

DETAILED DESCRIPTION:
Probiotic are live microorganisms that grant health effects to the host if consumed in sufficient amounts. Probiotic bacteria, which beneficially affect the host by improving the intestinal microbial balance, may affect the immune response, thus boosting the body system to combat against diseases.

Vaginal candidiasis can occur randomly in pregnant women. Vaginitis has been considered as one of the most common gynaecological condition affecting women worldwide. The prevalence of vaginitis was reported to be varied from 5% to 50% among different study populations across major continents such as the United States of America, Europe and South Asia. Vaginal candidiasis is one of the most common gynecological problems seen in primary care with Candida albicans account for 90% of the infection. The over-growth of this fungus in the vagina leads to a burning sensation in the vagina vulva, the production of heavy white/yellow curd-like discharge and/or an itchy vulva, pruritus, dyspareunia, dysuria, irritation, soreness of the vulva and other discomforting symptoms that will ensure frequent hospital visits.

During the past several decades, the many published surveys of vaginal flora specimens obtained from asymptomatic women have clearly shown that C. albicans may be present without the typical symptoms of yeast vaginitis. Moreover, the majority of women who have vaginal yeast also carry the organism in the gut. The typical rate of yeast carriage varies among populations and increases both after puberty and during pregnancy, which suggests an important role for pregnancy in cases of vaginal candidiasis. Probiotics are preferred compared to antibacterial drugs, such as clindamycin and metronidazole used for bacterial vaginosis treatment due to infection recurrence and drug resistance. It is a main concern that overuse of antibiotics could result in the development of antibiotic-resistant bacteria. Therefore, it is vital to find other alternatives to treat vaginal infections.

STP4 is manufactured under a HACCP and ISO 22000 certified manufacturing plant. The HACCP Codex Alimentarius is applied for the production of powdered Probiotics and Lactic Acid Bacteria used as food ingredients and the production of probiotics fermented solution used as food ingredients. The manufacturing plant also has been certified by Taiwan Quality Food (TQF) Scheme which they have met the requirement by Food Industry Research and Development Institute with the scope of processing of Ambient stable products. STP4 does not contain any porcine or bovine ingredients and has obtained the HALAL certification from Taiwan Halal Integrity Development Association (THIDA), Taiwan, which is recognized by JAKIM, Malaysia. STP4 capsules several strains of lactobacilli. The strains are Lactobacillus plantarum LP115, Lactobacillus helveticus LA25, Lactobacillus rhamnosus LRH10, Lactobacillus paracasei LPC12, Lactobacillus fermentum LF26, and Lactobacillus delbrueckii subsp. lactis LDL114. One capsule contains not less than 9.5 CFU of lactobacilli. The other ingredients are maltodextrin added with the ingredients and capsule shell made of hydroxypropyl methylcellulose.

A total number of 80 pregnant women (second and third trimester pregnancy) will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* 14-32 weeks pregnancy
* Confirmed vaginal candidiasis
* Positive vaginal yeast culture
* Willing to commit throughout the experiment

Exclusion Criteria:

* Self-declared illness that may have a potential to establish "leaky gut"
* Type-1 diabetes
* Long term medication (6 months or more) due to certain severe illness
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Second and third trimester pregnancy
Enrollment: 80 (Actual)
Dates: Start 2019-06-16 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2020-10-03 (Actual)

PRIMARY OUTCOMES:
To evaluate STP4 in reducing frequency of vaginal candidiasis re-occurring in pregnant women | 8 weeks
  To determine if oral administration of STP4 at 10 log CFU/day could reduce frequency (number and duration of times), of reoccurrence of vaginal candidiasis in pregnant women for 8-weeks compared to placebo

SECONDARY OUTCOMES:
To assess frequency of clinical symptoms | 8 weeks
  To determine if oral administration of STP4 at 10 log CFU/day could reduce frequency (number and duration of times) of clinical symptoms as assessed via questionnaire on vaginal candidiasis in pregnant women for 8-weeks compared to placebo. Questionnaire used is the Vulvovaginal Symptom Questionnaire (VSQ). Each of the 21 questions is answered as yes or no. Each yes carries 1 mark. A higher total score represents increase vulvovaginal symptom bother.
To assess concentrations of vaginal and cervical swab, cervico vaginal lavages fluid (CVL), and fecal samples | 8 weeks
  Concentrations include microbiota compositions, concentrations of cytokines and gene expressions of vaginal and cervical swab, cervico vaginal lavages fluid (CVL), and fecal samples of pregnant women on STP4 and placebo
To assess frequency in gastrointestinal symptoms | 8 weeks
  To determine if oral administration of STP4 at 10 log CFU/day could reduce frequency (number and duration of times), of gastrointestinal symptoms as assessed via questionnaire in pregnant women with candidiasis for 8-weeks compared to placebo
To determine health parameters of women and infants post-delivery | 12 months
  Parameters include health profiles of women and infants post-delivery as assessed via standard hospital medical records, from pregnant women on STP4 and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Fadlina Adnan, MD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- School of Industrial Technology, Universiti Sains Malaysia, Pulau Pinang, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No
Confidential

REFERENCES:
- [Derived] Ang XY, Roslan NS, Ahmad N, Yusof SM, Abdullah N, Nik Ab Rahman NN, Woon JJ, Teh CS, Todorov SD, Liu G, Liong MT. Lactobacillus probiotics restore vaginal and gut microbiota of pregnant women with vaginal candidiasis. Benef Microbes. 2023 Nov 23;14(5):421-431. doi: 10.1163/18762891-20220103. PMID 38350486